CLINICAL TRIAL: NCT00088270
Title: A Randomized, Open Label, Phase II Study of OSI-7904L Versus 5-FU/LV as First-Line Treatment in Patients With Unresectable, Locally Advanced or Metastatic Adenocarcinoma of the Biliary Tract
Brief Title: A Study of OSI-7904L Versus 5-FU/LV as Treatment in Patients With Biliary Tract Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: OSI Pharmaceuticals (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OSI-904-202
Record Dates: First submitted 2004-07-23; First posted 2004-07-26 (Estimated); Last update posted 2006-02-22 (Estimated); Status verified 2004-05

CONDITIONS: Locally Advanced or Metastatic Adenoca of the Biliary Tract
MeSH Terms: interventions — ((S)-2-(5-(1,2-dihydro-3-methyl-1-oxobenzo(f)-quinazoline-9-yl)methyl)amino-1-oxo-2-isoindolynyl)-glutaric acid; Fluorouracil; Leucovorin

INTERVENTIONS:
Drug: OSI-7904L
Drug: 5-Fluorouracil/Leucovorin

SUMMARY:
Multi-center, randomized Phase II study to evaluate the efficacy and safety of OSI-7904Lversus 5 FU/LV in biliary tract cancer.

ELIGIBILITY:
Inclusion Criteria:

Documented locally advanced or metastatic adenocarcinoma of the biliary tract; Adequate bone marrow, hepatic and renal function; Bilirubin <= 1.5 times the upper limit of normal; Age 18 years or older; Predicted life expectancy 12 weeks or more; Prior surgery and radiation therapy permitted provided patient has recovered adequately; At least 1 target lesion >= 20 mm (or >= 10 mm on spiral CT-scan); ECOG Performance Status 0-2; No prior chemotherapy for locally advanced or metastatic disease. Adjuvant/neo-adjuvant permitted if therapy was completed at least 12 months prior to study entry;

Exclusion Criteria:

Concurrent anticancer therapy while on study; History of other malignancy within the past 3 years except basal or squamous cell carcinoma or in situ cervical cancer; Symptomatic brain metastases which are not stable or have required radiation in the past 28 days;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58
Dates: Start 2004-08; Study Completion 2005-08

CONTACTS AND LOCATIONS:
Locations (21):
- United States (6):
  - Robert H. Lurie Comp. Cancer Ctr of Northwestern University, Chicago, Illinois
  - Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland
  - University of Michigan, Ann Arbor, Michigan
  - Wayne State University, Detroit, Michigan
  - Division of Hematology/Oncology, Columbus, Ohio
  - Vanderbilt Cancer Center, Nashville, Tennessee
- Belgium (3):
  - Institute Jules Bordet, 1000 Brussels
  - Dept Internal Medicine Gastrointestinal Oncology Unit, B-3000 Leuven
  - Department of Gastroenterology and GI Oncology, Brussels
- Germany (6):
  - Universitätsklinikum Charite Campus Virchow, 13353 Berlin
  - Allgemeines Krankenhaus St. Georg, 20099 Hamburg
  - Klinikum der J. W. Groethe-Universitat, 60590 Frankfurt
  - Innere Medizin Universitatsklinikum Heidelberg, 69115 Heidelberg
  - Medizinische Klinik II LMU-Klinikum-Großhadern, 81377 München
  - Tumorforschung Innere Medizinische Klinik, Essen
- Poland (2):
  - Klinika Nowotworow Gornego Odcinka, 02-791 Warszawa
  - Klinika Chemioterapii, 31-115 Krakow
- Romania (2):
  - Institutul Clinic Fundeni, 72437 Bucuresti
  - Oncology Institute Ion Chiricuta, Cluj-Napoca
- Switzerland (2):
  - Oncosurgery University Hospital of Geneva, 1211 Geneva 14
  - Multidisciplinary Oncology Center University Hospital CHUV, Lausanne